CLINICAL TRIAL: NCT05908812
Title: Relationship Between Parameters of Glycemic Control and Irisin Levels in Patients With Diabetes Mellitus Type 2 and Sarcopenic Obesity or Non-sarcopenic Obesity
Brief Title: Relationship Between Glycemic Control and Irisin in Type 2 Diabetic Patients With Sarcopenic or Non-sarcopenic Obesity
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Other Study IDs: 0023237|08/03/2023
Record Dates: First submitted 2023-04-18; First posted 2023-06-18 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Sarcopenia; Obesity; Diabetes Mellitus, Type 2
Keywords: Irisin protein; Hand Strength [E01.370.600.425.500]; Glycated Hemoglobin [D23.946.381.625.500.250]
MeSH Terms: conditions — Sarcopenia; Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Venous blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenic obesity: BMI>30, bioelectric impedance positive for sarcopenic obesity (FM% [fat mass percentage] female >43%, male >31% AND SMM/W [skeletal muscle mass/weight] female <28%, male <37%), any one of the physical performance test positive (5-times chair stand test >17 s OR handgrip strength test <35,5 kg for males, <20 kg for females).
- Non-sarcopenic obesity: BMI>30, bioelectric impedance negative for sarcopenic obesity.

SUMMARY:
The goal of this observational study is to compare glycemic control and irisin levels in subjects with diabetes mellitus type 2 with sarcopenic obesity vs non-sarcopenic obesity.

The main questions it aims to answer are:

Is glycemic control worse in diabetic patients with sarcopenic obesity? Are irisin levels higher in patients with non-sarcopenic obesity?

Participants will be asked to:

* Fill in three questionaries on lifestyle
* Perform two physical performance tests

The investigators will collect the following data:

* Anthropometric measurements
* Body composition by bioelectrical impedance analysis.
* Results of routine blood analyses
* Irisin levels by drawing a vial of blood from the antecubital vein

DETAILED DESCRIPTION:
Patients will be enrolled from our Diabetology Center. Eligible patients will be contacted by phone to be informed of the procedures and to schedule the visit.

The patients will come to the visit bringing the blood analyses they usually bring for the routine diabetologic visit; they will also be fasting for at least 3 hours, and abstaining from smoking and physical activity since the day before. All visits will be performed in the afternoon, at about 4-6 p.m.

Participants will be asked to:

* Fill in three questionaries (SARC-F [Strength, assistance with walking, rising from a chair, climbing stairs, and falls questionnaire], IPAQ-EIT [International Physical Activity Questionnaire validated in the Elderly Italian population], MEDI-LITE [Adherence to the Mediterranean diet questionnaire])
* Perform two physical performance tests (5-times chair stand test and handgrip test).

Anthropometric measurements will be assessed; body composition will be evaluated by bioelectrical impedance analysis. A venous blood draw will be executed for evaluation of irisin levels after signing a written consent form.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus type 2 diagnosed less than 10 years before
* age >60 years
* BMI (Body Mass Index) >30 kg/m2
* eGFR (estimated Glomerular Filtration Rate) >30 ml/min
* On stable antidiabetic therapy for at least 3 months

Exclusion Criteria:

* Insulin or insulin secretagogues use
* Diabetes mellitus type 1, previous diabetic ketoacidosis
* Neuromuscular diseases
* Endocrinopathies that may cause myopathies (hypercortisolism, GH [growth hormone] deficiency, acromegaly, adrenal insufficiency, partial hypopituitarism or panhypopituitarism, male hypogonadism, hyperparathyroidism, hypoparathyroidism)
* Severe vit. D deficiency (<12 ng/ml)
* Hemoglobinopathies
* Prolonged immobilization
* Pathologies with fluid retention (heart failure with NYHA [New York Heart Association] class III/IV, severe renal insufficiency, hepatic insufficiency)
* Active tumors in the past 5 years
* Severe arthritis of the knee or hip
* Pacemaker wearer

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected from our Center's patients. A physician will screen the eligible patients from the automatic search on the database from the program Smart Digital Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Differences in glycated hemoglobin and/or insulin resistance in diabetic patients with non-sarcopenic obesity vs patients with sarcopenic obesity | Baseline
  Differences in glycated hemoglobin or in HOMA-IR (Homeostatic Model Assessment for Insulin Resistance) in patients with sarcopenic obesity vs non-sarcopenic obesity

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Giorgino, MD, PhD, Principal Investigator — Director of U.O.C. Endocrinology and Metabolism, Policlinico di Bari
Locations (1):
- Policlinico di Bari, Bari, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Donini LM, Busetto L, Bischoff SC, Cederholm T, Ballesteros-Pomar MD, Batsis JA, Bauer JM, Boirie Y, Cruz-Jentoft AJ, Dicker D, Frara S, Fruhbeck G, Genton L, Gepner Y, Giustina A, Gonzalez MC, Han HS, Heymsfield SB, Higashiguchi T, Laviano A, Lenzi A, Nyulasi I, Parrinello E, Poggiogalle E, Prado CM, Salvador J, Rolland Y, Santini F, Serlie MJ, Shi H, Sieber CC, Siervo M, Vettor R, Villareal DT, Volkert D, Yu J, Zamboni M, Barazzoni R. Definition and Diagnostic Criteria for Sarcopenic Obesity: ESPEN and EASO Consensus Statement. Obes Facts. 2022;15(3):321-335. doi: 10.1159/000521241. Epub 2022 Feb 23. PMID 35196654
- [Result] Shoukry A, Shalaby SM, El-Arabi Bdeer S, Mahmoud AA, Mousa MM, Khalifa A. Circulating serum irisin levels in obesity and type 2 diabetes mellitus. IUBMB Life. 2016 Jul;68(7):544-56. doi: 10.1002/iub.1511. Epub 2016 May 24. PMID 27220658
- [Result] Oguz A, Sahin M, Tuzun D, Kurutas EB, Ulgen C, Bozkus O, Gul K. Irisin is a predictor of sarcopenic obesity in type 2 diabetes mellitus: A cross-sectional study. Medicine (Baltimore). 2021 Jul 2;100(26):e26529. doi: 10.1097/MD.0000000000026529. PMID 34190188

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/12/NCT05908812/Prot_ICF_000.pdf